CLINICAL TRIAL: NCT03503032
Title: Fenestrated Vs Non Fenestrated Extra-Cardiac Total Cavo-pulmonary Connection in Patients With Standard Preoperative Risk Profiles, A Prospective Randomized Study
Brief Title: Clinical Outcomes in Fenestrated Extra-Cardiac Fontan in Low Preoperative Risk Profiles
Status: Completed | Type: Observational
Sponsor: King Faisal Specialist Hospital & Research Center (Other)
Responsible Party: Sponsor
Other Study IDs: 1
Record Dates: First submitted 2018-04-09; First posted 2018-04-19 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Fontan Procedure
Keywords: Extracardiac Fontan; Total cavo-pulmonary connection; Fenestrated; Congenital heart defects; Pediatrics
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Fenestrated: Standard extracardiac fontan undergoing Fontan fenestration creation
  Interventions: Procedure: Extracardiac Fontan; Procedure: Fontan fenestration
- Non fenestrated: Standard extracardiac fontan without fenestration
  Interventions: Procedure: Extracardiac Fontan

INTERVENTIONS:
Procedure: Extracardiac Fontan — Extracardiac Fontan (Total cavo-pulmonary connection) will be constructed with a tube graft from the inferior vena cava to the pulmonary artery [applied to both arms]
  Other Names: Extracardiac Total cavo-pulmonary connection
Procedure: Fontan fenestration — Fontan fenestration created as a single 3 to 6mm communication between fontan channel and pulmonary venous atrium [Fenestrated arm]
  Groups: Fenestrated

SUMMARY:
Evaluation of fenestration benefit in Extra-cardiac total cavo-pulmonary connection (Fontan procedure) in single ventricle anomaly, comparing clinical outcomes of patients with low preoperative risk profiles in prospective study

DETAILED DESCRIPTION:
Study Population:

This study will include all patients referred for an elective Fontan procedure at the period of the study, who demonstrated a standard risk profile. An Informed consent will be obtained from the guardians before enrollment in the investigation. All procedures followed will be in accordance with institutional guidelines.

Randomization Technique:

Patients will be assigned to undergo either a fenestrated or non-fenestrated Extra-cardiac Fontan, based on a table of randomly generated numbers. Preoperative clinical data will be collected and compared to ensure appropriate randomization.

Preoperative Evaluation:

Enrolment Criteria:

Preoperative evaluation consists of ECG, transthoracic echocardiogram, and complete cardiac catheterization.

Patients with the following parameters will be eligible for enrollment in the study:

Sinus Rhythm Atriovnetricular valve regurgitation not more than mild Aortic (neoaortic) valve regurgitation not more than mild Normal systolic dominant ventricle function Mean pulmonary artery pressure not more than 15 mmHg (measured directly or estimated by pulmonary vein wedge pressure) Pulmonary vascular resistance not more than 2 woods unit End diastolic ventricular filling pressure not more than 8 mm Hg

Patient with the following will not be eligible for inclusion:

Patients with pulmonary artery distortion, stenosis or thrombus requiring surgical or interventional additional procedures before or during the Fontan operation. Pacemaker insertion before or during Fontan operation. Significant pulmonary arteriovenous malformations (AVMs) rendering fenestration potentially a cause of excessive cyanosis. Patients for whom the cardiology/cardiac surgery case conference decision is strongly in favor of fenestration for any other cause.

Ventricular filling pressure will be directly measured as the end-diastolic pressure in the dominant systemic ventricle. The degree of systemic atrioventricular valve regurgitation will be assessed semi-quantitatively by echocardiographic color Doppler, primarily based on width of jet origin. The regurgitation jet will be graded as none, mild, moderate, or severe. Rhythm is assessed with preoperative ECG or Holter monitor (if required). Coil occlusion of aortopulmonary collaterals is not an exclusion criterion and is recommended before the Fontan operation.

Operative Technique and postoperative management:

Treatment Patients underwent an extracardiac Fontan operation. The extracardiac Fontan channel will be constructed with a Polytetrafluoroethylene (PTFE) tube graft from the inferior vena cava to the pulmonary artery. The size if the graft is determined by the surgeon and ranged from 16 to 22 mm in diameter. The fenestration consists of a single 3- to 6-mm communication between the Fontan channel and the common atrium.

Postoperative treatment will include administration of captopril, and aggressive use of diuretics. All patients will receive aspirin (81 mg per day) and warfarin with a target International Normalized Ration INR of 2-2.5 beginning on the first postoperative day. To maximize caloric intake, patients ill not be fluid restricted after the initial postoperative period. All patients will be placed on fat free diet for 6 weeks. Chest tubes will be left in place until drainage is less than 5 mL/kg in a 24-hour period. A chest tube will be reinserted only if a symptomatic pleural effusion is diagnosed. Steroids and Octreotide will be started after 2 weeks of persistent drainage or immediately if Chylothorax is diagnosed biochemically.

The attending cardiologist and surgeon determined the need for and timing of postoperative cardiac catheterization. Patients will be discharged from the intensive care unit when hemodynamic and respiratory stability is ensured and a stable heart rhythm is maintained. The patients will be discharged from hospital after all chest tubes are removed and when the clinical status permits.

Assessment of Outcomes:

The primary end is the total length of chest tube drainage in days. If chest tube reinsertion is required during the same admission, this time will be added to the primary outcome. Other outcome variables include length of stay in the intensive care unit, total hospital stay in days, total amount of chest tube drainage, occurrence of stroke,readmissions, reoperation, or death within 90 days of discharge. All end points are defined a priori. The day of surgery counted as day 1 for all variables. All reoperations will be assessed including returning to the operating room for bleeding or poor hemodynamics, replacement of chest tubes, cardiac catheterization, and late fenestration.

Statistical Analysis:

Sample size estimates is based on a retrospective analysis of the last 100 patients who underwent the Fontan procedure at out institutionwith 80% power to avoid a type II statistical error. A reduction in total chest tube drainage days of 15% is considered clinically significant. The median length of chest tube drainage (estimated as one day less than the median postoperative length of hospitalization) was 19 days. Given a clinically significant difference of 15%, the calculated days of difference were 19 X 0.15 = 2.85. We set the relevant difference to be 3 days. Using a modified Lehr's equation for sample size in count data, we estimate the number in each group to be, n=4/〖(√(γ_1 )-√(γ_2 ))〗^2 =4/〖(√19-√16)〗^2 =31patients.

Descriptive statistics will be calculated for all variables. Medians and ranges describe continuous variables. Categorical variables will be summarized as frequencies. The Mann Whitney U test will be used for all continuous variables; analysis and Fisher's exact test will be applied for all dichotomous variables.

Count data for hospital length of stay, intensive care unit length of stay, and length of chest tube drainage will be compared by means of Poisson regression or Cox proportional hazards models. A probability value of 0.05 will indicate statistical significance. All calculations were performed with R-project statistical software (www.r-project.org).

ELIGIBILITY:
Inclusion Criteria:

* This study will includeall patients referred for an elective TCPC procedure at the period of the study, who demonstrated a standard risk profile
* Preoperative evaluation consisted of ECG, transthoracic echocardiogram, and complete cardiac catheterization.

Patients with the following parameters will be eligible for enrollment in the study:

* Sinus Rhythm
* Atriovnetricular valve regurgitation not more than mild
* Aortic (neoaortic) valve regurgitation not more than mild
* Normal systolic dominant ventricle function
* Mean pulmonary artery pressure not more than 15 mmHg (measured directly or estimated by pulmonary vein wedge pressure)
* Pulmonary vascular resistance not more than 2 woods unit
* End diastolic ventricular filling pressure not more than 8 mm Hg

Patient with the following will not be eligible for inclusion:

* Patients with pulmonary artery distortion, stenosis or thrombus requiring surgical or interventional additional procedures before or during the Fontan operation.
* Pacemaker insertion before or during Fontan operation.
* Significant pulmonary arteriovenous malformations (AVMs) rendering fenestration potentially a cause of excessive cyanosis.
* Patients for whom the cardiology/cardiac surgery case conference decision is strongly in favor of fenestration for any other cause.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients referred to King Faisal Specialist Hospital and Research Center in Jeddah for an elective (Fontan) Total cavopulmonar connection procedure at the period of the study, who demonstrated a standard risk profile.
Sampling Method: Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-04-12 (Actual); Study Completion 2023-04-12 (Actual)

PRIMARY OUTCOMES:
Duration of chest tube drainage | through study completion, an average of 1 year
  Total duration of days patient has been having chest tube inserted in his pleural cavities

SECONDARY OUTCOMES:
Length of hospital stay | through study completion, an average of 1 year
  Total duration of days patient spent in the hospital
Length of intensive care unit stay | through study completion, an average of 1 year
  Total duration of days patient needed to stay in intensive care unit
Total amount of chest tube drainage | through study completion, an average of 1 year
  Total amount of chest tube drainage throughout his post operative period in ml
Number of additional procedures | through study completion, an average of 1 year
  Any additional procedures were required in the postoperative period
Stroke | through study completion, an average of 1 year
  Any post operative cerebrovascular event
Readmissions | through study completion, an average of 1 year
  Number of readmissions to the hospital within 30 days of discharge
Death | Post operation and through 90 days of discharge from hospital
  Death post operation and through 90 days of discharge

CONTACTS AND LOCATIONS:
Overall Officials: Abdulbadee Bogis, MD, Principal Investigator — King Faisal Specialist Hospital & Research Center
Locations (1):
- KFSHRC, Jeddah, Westren, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Fontan F, Baudet E. Surgical repair of tricuspid atresia. Thorax. 1971 May;26(3):240-8. doi: 10.1136/thx.26.3.240. PMID 5089489
- [Background] de Leval MR, Kilner P, Gewillig M, Bull C. Total cavopulmonary connection: a logical alternative to atriopulmonary connection for complex Fontan operations. Experimental studies and early clinical experience. J Thorac Cardiovasc Surg. 1988 Nov;96(5):682-95. PMID 3184963
- [Background] Amodeo A, Galletti L, Marianeschi S, Picardo S, Giannico S, Di Renzi P, Marcelletti C. Extracardiac Fontan operation for complex cardiac anomalies: seven years' experience. J Thorac Cardiovasc Surg. 1997 Dec;114(6):1020-30; discussion 1030-1. doi: 10.1016/S0022-5223(97)70016-3. PMID 9434697
- [Background] d'Udekem Y, Iyengar AJ, Cochrane AD, Grigg LE, Ramsay JM, Wheaton GR, Penny DJ, Brizard CP. The Fontan procedure: contemporary techniques have improved long-term outcomes. Circulation. 2007 Sep 11;116(11 Suppl):I157-64. doi: 10.1161/CIRCULATIONAHA.106.676445. PMID 17846297
- [Background] Bando K, Turrentine MW, Park HJ, Sharp TG, Scavo V, Brown JW. Evolution of the Fontan procedure in a single center. Ann Thorac Surg. 2000 Jun;69(6):1873-9. doi: 10.1016/s0003-4975(00)01316-3. PMID 10892940
- [Background] Azakie A, Russell JL, McCrindle BW, Van Arsdell GS, Benson LN, Coles JG, Williams WG. Anatomic repair of anomalous left coronary artery from the pulmonary artery by aortic reimplantation: early survival, patterns of ventricular recovery and late outcome. Ann Thorac Surg. 2003 May;75(5):1535-41. doi: 10.1016/s0003-4975(02)04822-1. PMID 12735576
- [Background] de Leval MR, Dubini G, Migliavacca F, Jalali H, Camporini G, Redington A, Pietrabissa R. Use of computational fluid dynamics in the design of surgical procedures: application to the study of competitive flows in cavo-pulmonary connections. J Thorac Cardiovasc Surg. 1996 Mar;111(3):502-13. doi: 10.1016/s0022-5223(96)70302-1. PMID 8601964
- [Background] Bridges ND, Lock JE, Castaneda AR. Baffle fenestration with subsequent transcatheter closure. Modification of the Fontan operation for patients at increased risk. Circulation. 1990 Nov;82(5):1681-9. doi: 10.1161/01.cir.82.5.1681. PMID 2225370
- [Background] Bridges ND, Mayer JE Jr, Lock JE, Jonas RA, Hanley FL, Keane JF, Perry SB, Castaneda AR. Effect of baffle fenestration on outcome of the modified Fontan operation. Circulation. 1992 Dec;86(6):1762-9. doi: 10.1161/01.cir.86.6.1762. PMID 1451248
- [Background] Hsu DT, Quaegebeur JM, Ing FF, Selber EJ, Lamour JM, Gersony WM. Outcome after the single-stage, nonfenestrated Fontan procedure. Circulation. 1997 Nov 4;96(9 Suppl):II-335-40. PMID 9386120
- [Background] Thompson LD, Petrossian E, McElhinney DB, Abrikosova NA, Moore P, Reddy VM, Hanley FL. Is it necessary to routinely fenestrate an extracardiac fontan? J Am Coll Cardiol. 1999 Aug;34(2):539-44. doi: 10.1016/s0735-1097(99)00228-4. PMID 10440170
- [Background] Airan B, Sharma R, Choudhary SK, Mohanty SR, Bhan A, Chowdhari UK, Juneja R, Kothari SS, Saxena A, Venugopal P. Univentricular repair: is routine fenestration justified? Ann Thorac Surg. 2000 Jun;69(6):1900-6. doi: 10.1016/s0003-4975(00)01247-9. PMID 10892944